CLINICAL TRIAL: NCT05220787
Title: Evaluation of Efficacy and Safety of Extended Cold Stored Apheresis Platelets Versus Conventional Apheresis Platelets in Cardiac Surgery Patients
Brief Title: Extended Cold Stored Apheresis Platelets in Cardiac Surgery Patients
Acronym: CHASE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Moritz Stolla, MD (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Moritz Stolla, MD, Director of Platelet Transfusion Research Laboratory (Stolla Lab); Associate Medical Direct, Transfusion Service Swedish Medical Center; Assistant Professor of Medicine, University of Washington, Bloodworks
Organization: Bloodworks (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-01
Record Dates: First submitted 2021-10-11; First posted 2022-02-02 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Hemorrhage; Platelets; Defect; Bleeding; Surgical Blood Loss
MeSH Terms: conditions — Hemorrhage; Blood Platelet Disorders; Blood Loss, Surgical

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned to 1 of 2 treatment groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cold stored platelets in 100% plasma stored for 10-14 days (Experimental): Cold stored apheresis platelets in 100% plasma stored for 10-14 days, maximum of up to three units (3x10^11/unit) from the start of surgery until 24 hours after the end of surgery
  Interventions: Biological: Cold stored platelets in 100% plasma stored for 10-14 days
- Room temperature stored platelets in 100% plasma stored for up to 7 days (Active Comparator): Room temperature stored platelets in 100% plasma stored for up to 7 days, maximum of up to three units (3x10^11/unit) from the start of surgery until 24 hours after the end of surgery
  Interventions: Biological: Room temperature stored platelets in 100% plasma stored for up to 7 days

INTERVENTIONS:
Biological: Cold stored platelets in 100% plasma stored for 10-14 days — Subjects will receive cold stored platelets from the start of surgery until 24 hours after the end of surgery
  Arms: Cold stored platelets in 100% plasma stored for 10-14 days
Biological: Room temperature stored platelets in 100% plasma stored for up to 7 days — Subjects will receive room temperature stored platelets from the start of surgery until 24 hours after the end of surgery
  Arms: Room temperature stored platelets in 100% plasma stored for up to 7 days

SUMMARY:
This trial is being performed to evaluate the feasibility of the study protocol and to test the efficacy and safety of platelets stored at cold conditions (1-6°C) in 100% plasma for 10-14 days (CSP) in cardiac surgery patients who are actively bleeding and require platelet transfusion.

DETAILED DESCRIPTION:
Cardiac surgery featuring cardiopulmonary bypass (CPB) has a detrimental effect on platelet function. Contact with foreign surfaces causes a transient platelet dysfunction. The bleeding time is prolonged for the time on bypass and reverts to normal approximately one hour after cardiac surgery in uncomplicated cases. Hemorrhage following cardiac surgery with CPB can cause surgical re-exploration and increased mortality. The overall risk for surgical re-exploration is between 2.5-5%. Patients who undergo re-exploration due to excessive bleeding have a 2-6 fold increased mortality compared with non-bleeding patients. Storage of platelets at 1-6°C has the advantage of potentially prolonging storage times while reducing bacterial contamination. Room-temperature storage has led to a 5 day storage time limit since bacterial growth and septic reactions increase rapidly after 5-7 days. CSP were the standard of care in the 1960-70s. CSP were abandoned when a reduced platelet survival was observed in platelet radiolabeling studies. Nevertheless, CSP may have several advantages over RSP in the study population including a state of pre-activation and therefore a potentially superior hemostatic function. A small pilot trial investigating CSP in cardiac surgery patients in Norway found a non-significant trend towards improved bleeding control with CSP transfusions. However, data evaluating the in vivo efficacy of CSP is limited in scale and quality with mixed results. The investigators and others have shown that CSP have a superior function compared with RSP in vitro and more data are needed to clarify the relative efficacy of CSP in vivo. The investigators hypothesize that 1) CSP are more effective than RSP at reducing blood loss and improving platelet function in subjects actively bleeding due to cardiac surgery with cardiopulmonary bypass (CPB), and that 2) CSP are safe and do not lead to increased risks relative to RSP.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject age is greater than or equal to 18 years of age.
* 2. Subject can speak and read English.
* 3. Subject weight is greater than 40 kg.
* 4. Subject is scheduled for redo, triple valve, or complex aortic cardiac surgery with cardiopulmonary bypass.
* 5. Subject has ability to comprehend and willingness to sign Informed Consent Form (ICF).
* 6. If female of childbearing potential, must have a negative pregnancy test and agree to use one of the following methods of contraception during the course of study participation: abstinence, intrauterine contraception device, hormonal method, or barrier method.
* 7. Subject agrees to not participate in another interventional study during study participation.
* 8. The clinical site can obtain both possible platelet products (CSP and RSP) as needed per the study protocol given the subject's anticipated surgery date.

Exclusion Criteria:

* 1. Subject has history of known repeated, severe transfusion reactions.
* 2. Subject requires washed products, volume reduced products, or products with additive solution.
* 3. Subject is planned to receive autologous or directed transfusions.
* 4. Subject has or is expected to require post-surgical ventricular assist device (VAD), hemodialysis, or extracorporeal membrane oxygenation (ECMO) within 24 hours of the Study Treatment Window.
* 5. Subject is thrombocytopenic (less than 100 x 103 platelets/μL) on most recent measurement.
* 6. Subject is pregnant or breastfeeding.
* 7. Subject is a prisoner
* 8. Subject has active infection.
* 9. Subject refuses blood products.
* 10. Subject has a history of unprovoked deep vein thrombosis (DVT) or unprovoked pulmonary embolism (PE).
* 11. Subject has previously been enrolled and received a study platelet transfusion.
* 12. Subject has known bleeding diathesis (hemophilia, Von Willebrand Disease, or others)
* 13. At discretion of subject's physician, Sub-Investigator (SI), or Principle Investigator (PI).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-21 (Actual); Primary Completion 2024-10-29 (Estimated); Study Completion 2024-10-29 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the recruitment and accrual into the study protocol. | 24 hours following end of cardiac surgery
  Number of subjects screened and enrolled into the study protocol.

SECONDARY OUTCOMES:
Total allogeneic blood units transfused (RBCs only, platelets only, plasma only, and composite of all three) | Start of surgery to 24 hours after surgery
  Number of units
Chest tube output volume | 24 hours after completion of surgery
  volume of chest tube output measured in milliliters.
Hemostatic agents administered | 24 hours after completion of surgery
  The total individual doses of hemostatic agents
Number of subjects requiring surgical re-exploration due to uncontrolled bleeding | 24 hours after completion of surgery
  binary
Number of subjects with evidence of new infection or sepsis | Through post-op day 3
  per protocol definition
Number of subjects with evidence of a thrombotic event | Through study completion, an average of 3 weeks.
  per protocol definition
Number of subjects with evidence of liver injury. | Through post-op day 3
  Maximum post-operative change from pre-surgical baseline within the first three days
Hospital free days | Post-op through day 28.
  Number of days out of the hospital.
ICU free days | Post-op through day 28.
  Number of days out of the ICU
Ventilator free days | post-op through day 28.
  Number of days not on a ventilator.
Mortality | Post-op through day 28.
  To evaluate mortality at 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Moritz Stolla, MD, Principal Investigator — Bloodworks Northwest
Locations (1):
- Swedish Medical Center - Cherry Hill, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No